CLINICAL TRIAL: NCT00178906
Title: Acoustical Properties of Speech as Indicators of Suicidal Risk
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 9956
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Depression
Keywords: depression; suicide; voice
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This project is focused on acoustical, sound, analysis of speech in order to identify vocal characteristics of speech that are associated with suicidality. Speech samples will be collected from four populations with different mental health status: suicidal, ideational suicidal, depressed and those in remission from depression, (the control group). Speech of subjects will be recorded during routine diagnostic interview sessions. The speech samples will be acoustically analyzed via digital computer algorithms. The acoustical differences among those groups will be determined based on the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age Range: 25 to 65 years of age
* Participants must be depressed or be in remission from depression (have a history of depression)

Exclusion Criteria:

* speech impediment
* intoxication at time of interview

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely suicidal depressed patients; non-suicidal depressed patients;
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 1999-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Shiavi, PhD, Principal Investigator — Vanderbilt University; Ronald M Salomon, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States